CLINICAL TRIAL: NCT06626490
Title: Prospective Follow-up of the Prevision Hip Stem With Comparison of Different Implant Variants
Acronym: PREMO
Status: Not yet recruiting | Type: Observational
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-23015
Record Dates: First submitted 2024-09-19; First posted 2024-10-03 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Revision Total Hip Arthroplasty; Periprosthetic Fracture of Hip
Keywords: Patient-reported outcomes; Clinical performance and safety; Total hip arthroplasty implantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Prevision Revision hip endoprosthesis stem implantation — The Prevision hip endoprosthetic stem is a femoral part of a hip joint endoprosthesis. The system provides cementless and cemented variants. Prevision hip stems are modular with a short proximal and longer distal component, or monobloc hip stems. Modular components are coupled via a Prevision specific conical connection with a torque wrench and a tension nut to apply a predefined torsional moment on the connection. The distal component of modular Prevision stems can be combined with locking screws for additional bone fixation.
  Both types, the monobloc and the modular, provide a 12/14 taper that serves as a connection for metal or ceramic prosthesis heads. Prevision hip stems are combined at the acetabulum with a cementless or cemented acetabular cup.

SUMMARY:
The study design is confirmative for non-inferiority of the functional outcome of the implants and is intended to examine the safety and performance of the Prevision hip stem. The study is an observational post-market clinical follow-up study, and the study sites chose the stem variant depending on their own routine and indication.

DETAILED DESCRIPTION:
Generally, the advantage of the Prevision implant family is that all implant variants can be implanted with basically the same instrumentation, which makes it easier to switch to another variant. All implant variants will be available at the study sites and switching between the variants in the study will be encouraged.

The aim of the study is to prove the non-inferiority of the OHS functional outcome after two years to the predecessor implant generation, and comparable revision hip stems. In addition, the patient groups treated with the different variants, and outcome of these subgroups will be descriptively compared.

ELIGIBILITY:
Inclusion Criteria:

* Revision hip arthroplasty patients treated with a Prevision hip stem
* Written patient informed consent
* Patients are able to attend at follow-up examinations

Exclusion Criteria:

* Patients < 18 years at surgery
* Pregnancy at implantation
* Patients held in a custodial setting
* Patients in a relationship of dependence on the sponsor, the clinic or the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with indication of a hip revision
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2032-06 (Estimated); Study Completion 2033-03 (Estimated)

PRIMARY OUTCOMES:
Functional outcome of the hip revision surgery | after two years
  Oxford Hip Score:The Oxford Hip Score (OHS) is a joint-specific, patient-reported outcome measure designed to assess disability in patients undergoing total hip replacement (THR)

SECONDARY OUTCOMES:
Kaplan-Meier survival | after two years
  Kaplan-Meier Analysis is a standard statistical method to describe the survival of human subjects or medical products over a defined time period. The revision-free survival rate is the performance indicator of the product under investigation and confirms the clinical outcome of the knee prosthesis. Information on survival of the implant will be collected until the last follow-up of the study patients took place.
  1. revision for any reason
  2. hip stem revision
  3. aseptic hip stem revision
EQ-5D-5L Quality of Life | visits after 2 and 5 years
  EQ-5D is a standardized 5-dimension 5-level measure of the health status and is developed by the EuroQol Group in order to have a simple and generic measure for clinical and economic assessment. Instructions for the user are directly included into the questionnaire and it consists of two pages. One cover five different dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression) and the other one the EQ visual Analogue Scale (EQ-VAS). The VAS scale records the self rated health status of the patient from the level "the worst health you can imagine" to "the best health you can imagine".
Complications | visits after 2 and 5 years
Patient satisfaction | visits after 2 and 5 years
  Patient reported four-scale evaluation:
  * very satisfied
  * satisfied
  * unsatisfied
  * very unsatisfied
Pain (VAS Score) | visits after 2 and 5 years
  VAS Pain at Rest:
  0-100, lower is better
  VAS Pain under load:
  0-100, lower is better
  Patients are asked to mark a point on the line that corresponds to their current level of pain. This mark is then measured and converted into a numerical value, usually between 0 and 10 or 0 and 100, where 0 indicates no pain and the highest value indicates the most severe pain
Radiology: Hip stem subsidence | visits after 2 and 5 years
  Hip stem subsidence in mm.
Qualitative radiologic assessment | visits after 2 and 5 years
  Fracture healing; if radiolucent line > 2 mm, resorption, hypertrophy, cyst

CONTACTS AND LOCATIONS:
Overall Officials: Henning Windhagen, Prof. Dr., Principal Investigator — Orthopädische Kliniken im Annastift, MHH
Locations (1):
- Orthopädische Kliniken im Annastift, MHH, Anna-von-Borries-Str. 1-7, Hanover, Germany